CLINICAL TRIAL: NCT01577134
Title: Personal Resources of Elderly People With Multimorbidity: Fortification of Effective Health Behaviour
Brief Title: Personal Resources of Elderly People With Multimorbidity
Acronym: PREFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Centre of Gerontology (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government); Freie Universität Berlin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01ET1001B
Record Dates: First submitted 2012-03-19; First posted 2012-04-13 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Multimorbidity
Keywords: multimorbidity; autonomy; older adults; physical activity; intervention; behavior change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention to enhance physical activity (Experimental): Participants in this arm have high motivation to be regularly physically active. Face-to-face group intervention includes behavior change techniques to enhance physical activity.
  Interventions: Behavioral: Social-cognitive resource intervention
- Active control intervention (Active Comparator): Face-to-face group intervention includes behavior change techniques to enhance volunteering and improve attitudes towards volunteering.
  Interventions: Behavioral: Social-cognitive resource intervention
- Passive control intervention (Other): Waiting-list control group, who receives all information (that the active groups got) via mail after completion of 8.5 months follow-up.
  Interventions: Behavioral: no intervention

INTERVENTIONS:
Behavioral: Social-cognitive resource intervention — Intervention group that receives a behavior change technique intervention to increase volitional strategies and physical activity.
  Arms: Intervention to enhance physical activity
Behavioral: Social-cognitive resource intervention — Active control group that receives a behavior change technique intervention to increase volitional strategies and volunteering.
  Arms: Active control intervention
Behavioral: no intervention — Passive control group that receives no intervention until the 8.5 months follow-up. Subsequently, they receive the information by mail the active groups received within the intervention.
  Arms: Passive control intervention

SUMMARY:
PREFER II aims at developing psychological targeted theory- and evidence-based intervention components, which support older people with multiple illnesses in performing more physical activity. Many studies provide evidence for the importance of physical activity as a central mediator of health. This means that determinants of physical activity such as personal resources constitute an ideal target for interventions.

Within PREFER II, particularly positive views on ageing, attitudes, self-efficacy, planning and self-monitoring will be targeted in the interventions. These factors are important both for motivating older people with multiple illnesses to change their health behaviors and to translate such motivation into behavior.

ELIGIBILITY:
Inclusion Criteria:

* 64 years or older
* community-residing

Exclusion Criteria:

* regularly exercising

Min Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Baseline, 6 weeks, 10 weeks, 8.5 months, 12 months

SECONDARY OUTCOMES:
Change in quality of Life | Baseline, 6 weeks, 10 weeks, 8.5 months, 12 months
Change in self-reported perceived autonomy | Baseline, 6 weeks, 10 weeks, 8.5 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Tesch-Römer, Prof. Dr., Study Chair — German Centre of Gerontology; Ralf Schwarzer, Prof. Dr., Study Chair — Freie Universität Berlin
Locations (1):
- German Centre of Gerontology, Berlin, Germany